CLINICAL TRIAL: NCT02519140
Title: Assessing How the Viscosity of Submucosal Gel Injections Helps With Endoscopic Mucosal Resections
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-05-06
Record Dates: First submitted 2014-08-17; First posted 2015-08-10 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer; Colon Cancer
Keywords: Gastric cancer; colon cancer; EMR; biopsy; bariatric surgery
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cook medical EMR Gel (Experimental): Prospective study involving excised human stomachs and colon harvested from sleeve gastrectomies and colectomies performed for benign or malignant disease.
  Different Cook submucosal injections of varying viscosities will be injected into different areas of the excised stomachs or colons.
  Data collected will involve lifting characteristics and dissection adequacy of the varying viscosities of gel.
  Interventions: Drug: Cook Medical EMR Gel

INTERVENTIONS:
Drug: Cook Medical EMR Gel — Cook Medical EMR Gel will be injected submucosally into ex-vivo gastric or colonic tissue specimens
  Other Names: Cook Medical EMR Gel will be injected submucosally

SUMMARY:
This is a study to determine how the viscosity (thickness) of an FDA approved gel affects the ease in which endoscopic mucosal resections (EMR) can be performed.

DETAILED DESCRIPTION:
This is a study to determine how the viscosity (thickness) of an FDA approved gel made by Cook medical affects the ease in which endoscopic mucosal resections (EMR) - a type of endoscopic surgery performed for localised cancer - can be performed when the gel is injected submucosally. The lifting characteristics of the gel will be assessed by height and diameter and ease with which the subsequent EMR dissection can be performed. These characteristics would be assessed on excised human stomachs and colon, which are harvested during routine sleeve gastrectomy surgeries or colectomies, in an ex-vivo manner.

ELIGIBILITY:
Inclusion Criteria:

* Pts undergoing sleeve gastrectomy
* Pts undergoing colectomy

Exclusion Criteria:

* Unable to give or understand consent
* All of the excised tissue will be needed for diagnostic purposes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Lift Efficacy | 1 hour
  Lifting characteristics which would be measured by height of the mucosa after submucosal gel injection.

SECONDARY OUTCOMES:
Dissection Adequacy | 1 hour
  Dissection adequacy which would be measured by time which the gel stays within the tissues. Anything less than one hour will be considered failure.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Sherwinter, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Chandrasekhara V, Sigmon JC Jr, Surti VC, Kochman ML. A novel gel provides durable submucosal cushion for endoscopic mucosal resection and endoscopic submucosal dissection. Surg Endosc. 2013 Aug;27(8):3039-42. doi: 10.1007/s00464-013-2813-y. Epub 2013 Feb 8. PMID 23392984